CLINICAL TRIAL: NCT05063708
Title: To Evaluate the Activity and the Efficacy of Traditional Swallowing Therapy (TST) Plus Neuromuscular Electrostimulation (NMES) vs TST Plus Sham- NMES in Multiple Sclerosis People With Dysphagia
Brief Title: Neuromuscular Electrostimulation in Multiple Sclerosis People With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE/PROG.809; No 2019/R -Multi/ 005 (Other Grant/Funding Number: Italian MS Society Research Foundation)
Record Dates: First submitted 2021-08-10; First posted 2021-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-04

CONDITIONS: Deglutition Disorders; Multiple Sclerosis
Keywords: Neuromuscular electrostimulation Multiple Sclerosis
MeSH Terms: conditions — Deglutition Disorders; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study is a randomised double blind controlled study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Traditional dysphagia therapy plus sham Neuromuscular electrostimulation (Sham Comparator): Traditional dysphagia therapy (TDT) involved orofacial, lingual, and laryngeal motor exercises and compensatory swallowing strategies included various modifications of head, neck, and body postures and adjustment of food/liquid temperature, viscosity, and volume. The choice of specific strategies was based on the FEES findings and the clinical swallowing examination. The rehabilitative treatment will be administered in the 8 centers taking part to the study. The electrodes in this "sham" group will be placed in the same positions as the active treatment, with a current between 3 and 5 mA (average of 3.5 mA) current unable to perform muscle contraction. Every MS patient will be received 16 sessions of TDT according to their degree of dysphagia, contemporary associated with Sham neuromuscular electrostimulation two 30-min treatment a day, separated by a rest period of at least 45 minutes for four consecutive days per week, within a period of 4 weeks
  Interventions: Device: Sham Comparator: Traditional dysphagia therapy plus sham Neuromuscular electrostimulation
- traditional dysphagia therapy plus Neuromuscular electrostimulation (Experimental): Every MS patient will be treated with traditional dysphagia therapy, associated with an active neuromuscular electrostimulation. The amplitude will be increased until the subject will feel a 'grabbing sensation' which corresponded to muscular contraction. This will be the amplitude used for the therapy. This process will be repeated for the second channel of the stimulator. The typical electrical stimulus is at 80 Hz and at 300 microsec, and it will be adapted to avoid annoying stimulus to the patients. During therapy, both channels will be active. Every MS patient will be received 16 sessions of traditional dysphagia therapy according to their degree of dysphagia, contemporary associated with neuromuscular electrostimulation , according to our previous experiences, two 30-min treatment a day, separated by a rest period of at least 45 minutes for four consecutive days per week, within a period of 4 weeks.
  Interventions: Device: Experimental: traditional dysphagia therapy plus Neuromuscular electrostimulation

INTERVENTIONS:
Device: Experimental: traditional dysphagia therapy plus Neuromuscular electrostimulation — In the present study, VitalStim equipment will be used (VitalStim Therapy; Chattanooga Group, Chattanooga, TN, USA). Therapists received additional training and information on NMES by an experienced laryngologist certified to use surface electrical stimulation.
  Other Names: traditional dysphagia therapy
  Arms: traditional dysphagia therapy plus Neuromuscular electrostimulation
Device: Sham Comparator: Traditional dysphagia therapy plus sham Neuromuscular electrostimulation — Therapists received additional training and information on NMES by an experienced laryngologist certified to use surface electrical stimulation. The training was given according to the manual of the manufacturer, the VitalStim certification course (http://www.vitalstim.com).
  Other Names: traditional dysphagia therapy
  Arms: Traditional dysphagia therapy plus sham Neuromuscular electrostimulation

SUMMARY:
Dysphagia is a disabling, life-threatening symptom that can cause death in Multiple Sclerosis people (pwMS) through aspiration pneumonia. Speech therapists use behavioural therapies (compensatory and rehabilitative) to alleviate such swallowing problems, with limited benefit. Compensatory strategies such as postural changes and changes in food consistency, have been found to be partially effective, especially in patients with mild dysphagia and may be ineffective in patients with more severe dysphagia. The rehabilitative strategies include "no swallow exercises" which aim to strengthen isolated muscles used in swallowing (such as tongue strengthening) and "swallowing exercises" that aim at strengthening all the muscles used in swallowing while executing a hard, effortful, or prolonged swallow. To date, no randomized clinical trials have shown that rehabilitative strategies are effective. Neuromuscular electrical stimulation (NMES), often referred to as electrical stimulation, was introduced as a novel therapy for dysphagia in the late 2001. The principles of NMES in the limb rehabilitation literature are well established. However published protocols applying NMES to swallowing function have shown mixed results in people with stroke and only one study was published on MS people. This will be a double blinded, randomized clinical trial (patients and research staff blinded) with two arms: standard speech therapy plus Active NMES vs speech therapy with Sham NMES. The aim of this study is to determine whether NMES added benefit to a therapy program comprised of standard swallowing exercises in dysphagic pwMS.

DETAILED DESCRIPTION:
Recent studies has shown that dysphagia in MS is more frequent than previously believed, the real prevalence ranging from 33 to 43%. Dysphagia is a disabling, life-threatening symptom that can cause death in MS people through aspiration pneumonia. Dysphagia has also been reported in about 17% of patients with low disability (EDSS score lower than 2.5) . These figures, which are based on clinical evaluations, are undoubtedly higher when the symptom is evaluated by means of instrumental investigations . According to the De Pauw study , permanent dysphagia emerges in mildly impaired patients (EDSS 2-3), and becomes increasingly common as disability worsens, reaching a prevalence of 65% in the most severely disabled subjects (EDSS 8-9). Thus, diagnosis in the early stages may play an important role in limiting the consequences of this dysfunction. However, as patients themselves sometimes underestimate this symptom, diagnosis must be supported, as recently described in the literature, by functional tests and instrumental evaluations. A specific questionnaire (DYMUS: Dysphagia in Multiple Sclerosis) was published and validated for the assessment of dysphagia in MS. Its good internal consistency and the feasibility of administration has made it a reliable means to detect dysphagia in MS. In particular it consents to distinguish dysphagia to solids from dysphagia to liquids. However, a more detailed and objective evaluation is needed to investigate specific deficits and to plan appropriate rehabilitation; the Fiberoptic Endoscopy Evaluation of Swallowing (FEES) may be used for this purpose. In the 20 years since these initial reports, the FEES has become a validated technique for the evaluation of pharyngeal swallowing. The swallowing disturbances in MS are characterized by impairment of the oral and pharyngeal phases. Abraham et al. found impairment of the upper oesophageal sphincter in 100% of a small MS population . Calcagno et al., using a mixed clinical and instrumental examination, subdivided their population into three groups according to the severity of dysphagia: severe, moderate and slight. Severe dysphagia group showed impairment of both oral and pharyngeal phases of swallowing, moderate dysphagia group showed motor impairment of the tongue, lips, velum or larynx, while the mild dysphagia group showed deficiency either of the velum or of the glottic closure. In the same paper, Calcagno et al. found that the compensatory strategies resolved dysphagia in about 94% of the cases (46 pts. Out of 49) These strategies help to redirect and improve the food flow, avoiding aspiration and reducing the risk of pneumonia, but patients remain dysphagic and always need to perform compensatory strategies. This seem to be the only study evaluating the rehabilitative approach, but it was not a control study. The role of food was highlighted in a recent paper showing that the main effect of food hardness is a delay in oral ejection time, which strongly delays total swallowing time, whereas pharyngeal bolus transit is dependent on its viscosity. Recently, a pilot study has shown as NMES could probably improve voice quality in MS patients: in fact, dysarthria has been proven to affect quality of life in MS patients .

NMES is a form of muscle stimulation with short electrical pulses that is frequently used in physiotherapy to strengthen healthy muscles and has been well described for several decades. NMES is used with a variety of different parameters for different types of treatment, since muscle contraction depends on different electrical parameters. An increase in frequency will result in an increased tension of the stimulated muscle, whereas increased intensity spreads current over a larger area, stimulating more motor units. Lastly, increasing the current duration causes more motor unit activation. NMES can be used for either muscle strengthening, retardation of atrophy or muscle re-education, and different stimulation parameters have to be chosen for each of these three applications of NMES. The use of NMES in dysphagia treatment is relatively new; the first study was published in 2001 . Although Logemann reported that the therapeutic effects of NMES still lacks convincing supporting evidence, several studies have been carried out Research using NMES, including randomized controlled trials, has demonstrated functionally improved swallowing with subjects moving from modified diets to more normal diet and fluids when NMES is used in conjunction with traditional therapy, but not when used in isolation .

Moreover, recent UK guidelines from the National Institute of Clinical Excellence (NICE) recognized the positive results from these trials and promoted a further research to support the routine clinical use. NMES has been used in a wide range of patients, suffering from diverse pathologies: from head and neck cancer, to post-stroke dysphagia, obtaining different results . Although it has been hypothesized, that neuromuscular electrical stimulation might enhance muscle strength in weak and disused oro-pharyngeal muscles, its clinical effectiveness remains unclear. Regardless the mechanism of action, clinical results showed that NMES enhances laryngeal elevation , reduces upper esophageal sphincter pressure and it enhances tongue base retraction during swallowing in health volunteers . As reported by Oh and Hamdy , the improvement of the swallowing function in stroke, after electrical stimulation is correlated with cortical reorganization, suggesting that multiple sessions of NEMS of the neck muscles could improve swallowing function also trough the recruitment of new cortical areas.

NMES has poor been used in treating dysphagia in MS patients A pilot study performed with pharyngeal electrical stimulation for dysphagia associated with MS showed an improvement in penetration and aspiration scale, suggesting a potential benefit for the treatment of this symptom.

However, this type of treatment can be performed only in specialized centers and it is probably more invasive than NMES. In 2009, Bogaardt conducted a Class IV trial with a sample of 25 patients with MS. The primary focus of the study was to examine the effects of NMES on pooling of saliva or liquid in the valleculae and pyriform sinuses. Six of the 25 patients had significant reduction in pooling of saliva in the pyriform sinuses, and 23 participants reported through a questionnaire that their swallowing had improved. This seem to be the unique paper focusing on the therapeutic effects of NMES in MS patients. Simonelli et al recently published about the use of NMES in people with stroke and dysphagia. The methodology resulted safe with a good effectiveness in add on with traditional speech therapy. In fact, combined treatment seem to reduce the risk of penetration and aspiration in stroke dysphagic people.

The aim of the study is to determine whether NMES added benefit to a therapy program comprised of standard swallowing exercises in dysphagic pwMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: definite MS (Thompson et al 2018)
* Stability: recruited subjects must be in a stable phase of the disease, without relapses which induce worsening > 1 point in the EDSS and with an EDSS <=8
* ASHA<6 and DYMUS >2
* Novelty: subjects should not have been trained with dysphagia program in the last 6 month
* Mini-Mental State Examination: > 24

Exclusion Criteria:

* Dysphagia related to other diseases
* Presence of tracheal cannula
* Local or general contraindications to the use of equipment for electrical muscle stimulation of the neck
* Malignancies or acute inflammation in the anterior region of the neck.
* Lack of collaboration due to mental impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
change from American Speech-Language Hearing Association (ASHA) score baseline at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at ASHA score between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent the primary outcome.ASHA suggests that patients should be divided in groups from level 1 (individuals cannot swallow anything safely by mouth) to level 7 (individual's ability to eat independently is not limited by swallowing function

SECONDARY OUTCOMES:
Change from Dysphagia in Multiple Sclerosis (DYMUS) scale at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at DYMUS score between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia. therapy plus neuromuscular electrostimulation will represent one of secondary outcome.It's a 10 item self administered questionnaire. The answer "yes" is a red flag for dysphagia
Change from Fiber-optic endoscopic evaluation of swallowing /Dysphagia at Outcome Severity Scale (FESS/DOSS score) at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at FESS/DOSS score between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent one of secondary outcome. FEES is scored using DOSS levels (scored from 7 to 1). In particular, level 7 is consistent with full oral nutrition with a normal diet
Change from Mini Nutritional Assessment at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at Mini Nutritional Assessment between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent one of secondary outcome. The score is from 0 to 30. The up score represents a normal value
Change from the Swallowing Quality of life questionnaire at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at the Swallowing Quality of life questionnaire between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent one of secondary outcome. The minimum and maximum score per subscale ranges from 0 to 100, indicating extremely impaired quality of life versus no impairment experienced by the individual
Change from Penetration and Aspiration Score at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at the Penetration and Aspiration Score between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent one of secondary outcome. The score is from 1 (no penetration) to 7 (severe aspiration)
Change from Pooling score at 12 weeks | after 16 sessions of treatment and after 12 weeks from the end of treatment
  The mean difference at Pooling score between group treated with traditional dysphagia therapy plus sham Neuromuscular electrostimulation vs group traditional dysphagia therapy plus neuromuscular electrostimulation will represent one of secondary outcome. The score is from 4 (no dysphagia) to 11 (severe dysphagia)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Grasso, MD, Principal Investigator — Fondazione Santa Lucia Rome Italy
Locations (1):
- Santa Lucia foundation, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Logemann JA. The effects of VitalStim on clinical and research thinking in dysphagia. Dysphagia. 2007 Jan;22(1):11-2. doi: 10.1007/s00455-006-9039-2. Epub 2007 Jan 10. No abstract available. PMID 17216392
- [Background] Simonelli M, Ruoppolo G, Iosa M, Morone G, Fusco A, Grasso MG, Gallo A, Paolucci S. A stimulus for eating. The use of neuromuscular transcutaneous electrical stimulation in patients affected by severe dysphagia after subacute stroke: A pilot randomized controlled trial. NeuroRehabilitation. 2019;44(1):103-110. doi: 10.3233/NRE-182526. PMID 30714980
- [Result] Alali D, Ballard K, Bogaardt H. Treatment Effects for Dysphagia in Adults with Multiple Sclerosis: A Systematic Review. Dysphagia. 2016 Oct;31(5):610-8. doi: 10.1007/s00455-016-9738-2. Epub 2016 Aug 4. PMID 27488370
- [Result] Bergamaschi R, Crivelli P, Rezzani C, Patti F, Solaro C, Rossi P, Restivo D, Maimone D, Romani A, Bastianello S, Tavazzi E, D'Amico E, Montomoli C, Cosi V. The DYMUS questionnaire for the assessment of dysphagia in multiple sclerosis. J Neurol Sci. 2008 Jun 15;269(1-2):49-53. doi: 10.1016/j.jns.2007.12.021. Epub 2008 Feb 15. PMID 18280504
- [Result] Ginocchio D, Alfonsi E, Mozzanica F, Accornero AR, Bergonzoni A, Chiarello G, De Luca N, Farneti D, Marilia S, Calcagno P, Turroni V, Schindler A. Cross-Cultural Adaptation and Validation of the Italian Version of SWAL-QOL. Dysphagia. 2016 Oct;31(5):626-34. doi: 10.1007/s00455-016-9720-z. Epub 2016 Jul 21. PMID 27444734
- See also: This platform is utilized by our institution for raw data — http://zenodo.org
- Available data/document: Analytic Code — http://zenodo.org
- Available data/document: Statistical Analysis Plan — http://zenodo.org

DOCUMENTS (1):
  • Study Protocol (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT05063708/Prot_000.pdf